CLINICAL TRIAL: NCT06008340
Title: Effect of Right Ventricle Lead Position on The Psychological Aspects of Patients With A Dual Chamber Pacemaker; A Prospective Comparative Controlled Study
Brief Title: Effect of Right Ventricle Lead Position on The Psychological Aspects of Patients With A Dual Chamber Pacemaker
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hassan El-Shirbiny, Principal investigator, Kafrelsheikh University
Other Study IDs: Pacing on Anxiety/ Depression
Record Dates: First submitted 2023-08-09; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Pacing-Induced Cardiomyopathy
Keywords: Anxiety; Depression; Psychological effect; Dual chamber; Pacemaker; Pacing
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dual chamber Pacemaker — Anti bradycardia device implanted in patients with complete heart block, the device has 2 leads, one in the RT atrium and the other in RV. The RV lead positioned either apical or septal

SUMMARY:
The purpose of the current study was to determine the factors associated with increased levels of anxiety and depression both before and after pacemaker implantation and examine if changes in these symptoms occur during the first postoperative year.

DETAILED DESCRIPTION:
Both clinical and experimental studies declared that RV pacing and the position of RV lead may lead to ventricular desynchrony, mimics that of LBBB with subsequent abnormal mechanical and electrical activation of the ventricles . This results in changes in cardiac perfusion, hemodynamics, metabolism and mechanical function .

With time, RV pacing may also lead to LV remodeling and structural changes . Also, it has been mentioned that the presence of mechanical desynchrony after long-term RV pacing especially the apical one is linked with reduced LV systolic function and deterioration in the functional capacity and psychological aspects of the patients also in some cases adverse clinical outcomes such as heart failure, atrial fibrillation and death However, in daily clinical practice, not all patients with RV apical pacing will have these adverse events.

Patients' depression and anxiety before and after pacemaker implantation have been understudied. National and international literature show only few studies about anxiety and depression in patients who experience a pacemaker but more research has reported that these two variables are heavily noticed in cardiovascular patients.

In fact, they are so frequent in patients with coronary artery disease, heart failure, and in patients who had an implanted defibrillator. It has been suggested that anxiety and depression have a prevalence ranging from 18% to 50% in cardiac patients . The few studies that have studied anxiety and depression in pacemaker patients researched these variables only in an unfaithful time from the implantation and without considering any changes before and after the pacemaker implantation.

In elderly population on the consequent increase of patients with pacemakers, this problem becomes an essential one to study to support healthcare providers to know not only the problem, but also who is at high risk to develop anxiety and depression. Research has illustrated that lower levels of anxiety and depression among elderly patients are linked with perceptions of higher quality of life and less need for the use of health services. The improvement of wellbeing in elderly patients has implications for health care providers designing preoperative and follow up care for patients undergoing pacemaker Implantation.

ELIGIBILITY:
Inclusion Criteria:

* implantation of a dual-chamber pacemaker,
* the ability to write and read the Arabic language,
* adequate follow-up and
* patients older than 18 years who were hospitalized for the first time for the implantation procedure

Exclusion Criteria:

* Patients with history of psychiatric illness (mental, emotional, or behavioral disorders),
* with a serious chronic disease,
* with implantable cardioverter defibrillator or biventricular pacemaker and
* patients who had not a stable programming of their device from the implantation.
* patients less than 18 years old,
* family and social environment problems prior and subsequent to PM implant,
* financial problems

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from heart block and indicated for permanent cardiac pacemaker implantation
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Lead position and anxiety/ depression | one year
  Assessment of the effect of the pacemaker lead position in the right ventricle on the psychological aspects of the patients in 1 year follow up period.

SECONDARY OUTCOMES:
Co morbidities and anxiety / depression | one year
  Assessment the correlation between hypertension, diabetes , ischemia and variable pacemaker complications on the anxiety and depression of the patients in 1 year follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Reda Baiomy, PHD, Study Director — Kafrelsheikh University
Locations (1):
- Kafrelsheikh university, Kafr ash Shaykh, Egypt

REFERENCES:
- [Background] Prinzen FW, Peschar M. Relation between the pacing induced sequence of activation and left ventricular pump function in animals. Pacing Clin Electrophysiol. 2002 Apr;25(4 Pt 1):484-98. doi: 10.1046/j.1460-9592.2002.00484.x. PMID 11991375
- [Background] Tops LF, Schalij MJ, Holman ER, van Erven L, van der Wall EE, Bax JJ. Right ventricular pacing can induce ventricular dyssynchrony in patients with atrial fibrillation after atrioventricular node ablation. J Am Coll Cardiol. 2006 Oct 17;48(8):1642-8. doi: 10.1016/j.jacc.2006.05.072. Epub 2006 Sep 27. PMID 17045901
- [Background] Polikandrioti M, Tzirogiannis K, Zyga S, Koutelekos I, Vasilopoulos G, Theofilou P, Panoutsopoulos G. Effect of anxiety and depression on the fatigue of patients with a permanent pacemaker. Arch Med Sci Atheroscler Dis. 2018 Feb 5;3:e8-e17. doi: 10.5114/amsad.2018.73231. eCollection 2018. PMID 30775584
- [Background] Chesney MA, Rosenman RH. Type A behavior: Observations on the past decade. Heart Lung. 1982 Jan-Feb;11(1):12-9. No abstract available. PMID 6915919